CLINICAL TRIAL: NCT00438685
Title: Development of Outpatient MST for Dually Diagnosed Youth
Brief Title: Outpatient Adolescent Treatment for Comorbid Substance Use and Internalizing Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Ashli J. Sheidow, MUSC
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21DA017118-01 (NIH); R21DA017118 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2010-07

CONDITIONS: Substance-Related Disorders; Depressive Disorder; Anxiety Disorder
Keywords: Substance-Related Disorders; Depressive Disorder; Anxiety Disorder; Adolescent; Behavior Therapy; Cognitive Therapy; Outpatients; Family Relations; Systems Theory
MeSH Terms: conditions — Substance-Related Disorders; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Outpatient MST/OPTION-A
Behavioral: Usual Services

SUMMARY:
Adolescent substance abuse results in significant negative outcomes and extraordinary costs for youths, their families, communities, and society. Moreover, rates of psychiatric comorbidity among substance abusing youth range from 25% up to 82%, and youths with a dual diagnosis have worse outcomes and are more than twice as costly to treat than their counterparts with no comorbidity. This project was a pilot test of a new treatment, OPTION-A, which was adapted from Multisystemic Therapist (MST) and other evidence-based interventions to specifically treat youth presenting for outpatient treatment of comorbid substance use and internalizing disorders. The project was a randomized controlled pilot trial comparing the experimental treatment to usual services in the community.

DETAILED DESCRIPTION:
Adolescent substance abuse results in significant negative outcomes and extraordinary costs for youths, their families, communities, and society. Moreover, rates of psychiatric comorbidity among substance abusing youth are high and youths with a dual diagnosis are more costly to treat. At the time of this study, however, no outpatient treatments had been tested specifically for treating youth with co-occurring substance use disorders and mental health diagnoses. The current project aimed to adapt and evaluate Multisystemic Therapy (MST), a well validated treatment for chronic behavioral problems or serious emotional disturbance in adolescents, to treat dually diagnosed youth using an outpatient model of service delivery.

A pilot trial was conducted with 40 dually diagnosed youth randomly assigned to treatment conditions, with 20 receiving the experimental treatment (OPTION-A) and 20 receiving usual outpatient services. Specific aims were:

Specific Aim 1: The primary aim of the present research was to adapt and test OPTION-A for use in outpatient settings to treat youth diagnosed with a substance use disorder and comorbid internalizing disorder. We hypothesized that youth receiving OPTION-A would exhibit significantly less drug use (e.g., youth self-reports and urine screens) than control youth who received usual services, and that youth receiving OPTION-A would exhibit significant improvement on indices of mental health (e.g., combined youth and caregiver reports on diagnostic interviews and youth, caregiver, and teacher reports of internalizing symptoms) compared to control youth Specific Aim 2: In addition to improved symptomatology, the current research aimed to test the effectiveness of OPTION-A to improve youth functioning in other domains pertinent to successful adolescent development. We hypothesized that youth receiving OPTION-A would evidence improved behavioral (e.g., youth, caregiver, and teacher reports of externalizing), school (e.g., school attendance), and family functioning (e.g., youth and caregiver reports of family adaptability and cohesion) compared to control youth who received usual services.

Specific Aim 3: The final aim of the proposed research was to provide services that are more acceptable to consumers than are usual services provided in the community. We hypothesized that youth and families receiving OPTION-A would experience significantly greater consumer satisfaction than control youth and families who received usual services.

ELIGIBILITY:
Inclusion Criteria:

* Presentation for outpatient treatment
* 12 to 17 years of age
* Youth residing with at least one adult caregiver who serves as a parent figure
* Substance Abuse or Dependence Disorder
* Axis I Internalizing Disorder (Mood Disorder or Anxiety Disorder), based on the Diagnostic Interview Schedule for Children (DISC-IV; Shaffer, Fisher, Lucas, Dulcan, & Schwab-Stone, 2000)

Exclusion Criteria:

* Pervasive Developmental Disorder
* Psychotic Disorder
* Severe or profound mental retardation (IQ of 45 or below)
* Families previously receiving Multisystemic Therapy

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2004-10; Primary Completion 2007-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Urine Drug Screen at 4 weeks, 8 weeks, 12 weeks, 24 weeks
Score on Depression/Anxiety Scale (RCADS) at 4 weeks, 8 weeks, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Measured at Intake, 3 Months, and 6 Months
Global assessment of symptoms
Parenting
School
Behavioral
Family relationship/communication/problem solving
Consumer satisfaction
Daily Drug/Alcohol use

CONTACTS AND LOCATIONS:
Overall Officials: Ashli J Sheidow, PhD, Principal Investigator — Medical University of South Carolina, Department of Psychiatry & Behavioral Sciences, Family Services Research Center; Scott W Henggeler, PhD, Study Chair — Medical University of South Carolina, Department of Psychiatry & Behavioral Sciences, Family Services Research Center
Locations (1):
- Medical University of South Carolina, Department of Psychiatry & Behavioral Sciences, Family Services Research Center, Charleston, South Carolina, United States